CLINICAL TRIAL: NCT04882722
Title: Opinion Survey on Postpartum Pelvic Floor Rehabilitation According to the Quality of Information Provided by the Health Care Providers
Brief Title: Postpartum Pelvic Floor Rehabilitation and Information Provided by the Health Care Providers
Acronym: PPFR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD21_0027
Record Dates: First submitted 2021-04-28; First posted 2021-05-12 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-04

CONDITIONS: Recovery of Function
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Self-questionnaire reported before the first PPFR session and after the last session

SUMMARY:
The aim of this work is to evaluate the experience of Postpartum Pelvic Floor Rehabilitation (PPFR) according to the information given by the health care providers. There is to improve medical practice and to give the right information in at the right time to the patient.

DETAILED DESCRIPTION:
Postpartum Pelvic Floor Rehabilitation is an important central stage of the postpartum period. It allows, if it is well done, to reduce complications related to childbirth, (pelvic floor disorders: urinary, sexual or anal disorders ) and to increase quality of life of women in postpartum period.

But, what about the woman's opinion and experience of PPFR? Previous studies have evaluated the effectiveness of PPFR but not the woman's experience.

It is interesting to evaluate the experience of PPFR according to the information given by the health care providers. There is to improve medical practice and to give the right information in at the right time to the women

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing postpartum pelvic floor rehabilitation at the Departmental Hospital Center of Vendee

Exclusion Criteria:

* Refusal to participate in the study
* Patient did not complete all her PPFR sessions at the Departmental Hospital Center of Vendee
* Patient unable to understand the protocol, read the information note and answer the questionnaires
* Patient under tutelage, curatorship, mandate of future protection, family habilitation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women undergoing pelvic floor rehabilitation at the Departmental Hospital Center of Vendee
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall experience of the PPFR according to information given by the health care providers | through study completion, an average of 5 weeks
  Self-evaluation of the overall experience of postpartum pelvic floor rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, Dr, Principal Investigator — Departmental Hospital Center of Vendee
Locations (1):
- Departmental Hospital Center of Vendee, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No